CLINICAL TRIAL: NCT06410482
Title: Comparison Between the Analgesic Efficacy of the Ultrasound Penile Block Versus Ultrasound Caudal Epidural for Pediatric Hypospadias Surgeries: A Prospective Randomized Double Blinded Trial
Brief Title: Analgesia in Pediatric Hypospadias Surgeries
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Esraa Gaafer, Resident Doctor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: pediatric hypospadias
Record Dates: First submitted 2023-11-14; First posted 2024-05-13 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: Hypospadias
MeSH Terms: conditions — Hypospadias

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- US guided caudal block Anesthesia (Experimental): Children will receive caudal block analgesia
  Interventions: Procedure: US guided caudal block
- Dorsal penile nerve block Anesthesia (Active Comparator): Children will receive Penile block analgesia
  Interventions: Procedure: Dorsal penile nerve block

INTERVENTIONS:
Procedure: US guided caudal block — After placing the patient in the left lateral position (hips and knees flexed) following monitoring and induction of anaesthesia, the field will be sterilized with 70% alcohol in 2% chlorhexidine.
  Initial scanning in the transverse plane allows for visualization of the midline and identification of the sacrococcygeal ligament between the 2 sacral cornua. The 2 cornua resemble the 2 eyes of a frog and thus are collectively called the frog-eye sign. The US probe is then rotated 90 degrees to acquire a longitudinal view. The needle is then advanced at a 20-degree angle with needle tip and length visualization Once the needle is confirmed to be in the caudal space on the screen, carefully aspirate to confirm absence of CSF or blood.
  A slow injection of the local anaesthetic can then be performed, dose of (0.2 mL/kg 0.25% bupivacaine and 1 μg/kg of dexmedetomidine
  Arms: US guided caudal block Anesthesia
Procedure: Dorsal penile nerve block — after general anesthesia induction. With the patient in the supine position. After skin sterilization the US linear probe will be transversely placed on the root of the penis. After placing the penis in gentle traction, a50 mm block needle will be inserted from the lateral part of the penis root towards the dorsal section of the penis with the in-plane technique, It will be advanced through Dartos fascia until resistance to the needle disappeared.
  Once the superficial sheath will be passed, the tip of the needle will be advanced into Buck's fascia and then positioned between Buck's fascia and tunica albuginea, lateral to the dorsal artery. After making sure there will be no blood with negative aspiration, half of the total 0.2 mL/kg dose of 0.25% bupivacaine will be administered while observing its distribution with US. The same procedure will be then repeated on the other side of the penis.
  Arms: Dorsal penile nerve block Anesthesia

SUMMARY:
The primary aim of the current study will be to use the duration until the first postoperative analgesic requirement after two different block techniques to compare the analgesic effect.

The secondary aims will be to compare the two methods for postoperative Children's Hospital Eastern Ontario Pain Scale (CHEOPS) scores, complications and parental satisfaction scores.

DETAILED DESCRIPTION:
Hypospadias, seen in every 200-300 births, is one of the most common congenital anomalies of the penis and is defined as the urethral meatus being located in the ventral part of the penis instead of its normal place.

Although current guidelines propose an optimal age for hypospadias repair of 6-18 months , patient ages vary widely, from infants to adults, in daily practice. According to the literature, hypospadias surgery can be performed in a wide age range of 6 months-12 years. The age of the patients undergoing hypospadias surgery in our country can vary between 1 and 10 years. The surgery of this anomaly is very painful in the postoperative period and requires long-term analgesia. Regional anesthesia methods combined with general anesthesia play an important role in providing effective and long-term postoperative pain control in pediatric penile surgery. These methods also reduce postoperative morbidity, enable early mobilization and significantly decrease the need for narcotic analgesics.

A dorsal penile nerve block (DPNB) and caudal epidural block (CEB) are commonly used regional anesthesia techniques for postoperative pain control in hypospadias repair. CEB is the more commonly used neuraxial block method for providing effective postoperative analgesia in lower abdominal, urogenital and lower extremity surgical operations in pediatric patients. However, it has recently been suggested in the literature that peripheral nerve blocks should be preferred to neuraxial blocks as they provide longer-term analgesia and have fewer side effects. DPNB is a peripheral nerve block method that has been widely used for various penile operations since it will be first defined in the mid-1970s. This method is mostly used with the landmark technique. It will be first used by Sandeman et al via the out-of-plane technique with ultrasound (US) and will be reported to provide effective analgesia in the postoperative period. Suleman et al described DPNB for the first time with the in-plane technique, indicating that the tissue and neurovascular structures of the penis could be better distinguished in the transverse plane in ultrasound (US). A limited number of studies have shown the technique to provide more effective and longer term postoperative analgesia compared to the landmark technique and CEB.

ELIGIBILITY:
Inclusion Criteria:

* • Children aged 1-7 years old

  * ASA I and II
  * Children scheduled for primary hypospadias repair

Exclusion Criteria:

* • Patient's guardian refusal to participate in the study.

  * Children with Behavioural changes; physical or developmental delay; neurological disorder or psychological disorder.
  * Children on sedative or anticonvulsant medication.
  * Bleeding diathesis
  * Infection of injecting area
  * significant organ dysfunction, cardiac, liver or mental retardation.
  * Congenital low back anomaly.
  * Known allergy to the study drugs

Ages: 1 Year to 7 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 26 (Estimated)
Dates: Start 2024-05 (Estimated); Primary Completion 2025-05 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
postoperative pain and analgesic requirement after two different block techniques to compare the analgesic effect. | 24 hours after the end of surgery
  Postoperative pain will be assessed using the Children's Hospital Eastern Ontario Pain Scale (CHEOPS) score at 30 minutes, 1, 2, 6, 12 and 24 hours.
  the minimum score is 4 (better outcome) and the maximum score is 13 (worse outcome). A score ≥ 5 should be considered sufficient to administer an analgesic to the child, where a score of ≥ 8 makes it a requirement to administer an analgesic to the child.

SECONDARY OUTCOMES:
Postoperative complications | 24 hours after the end of surgery
  Postoperative complications as nausea, vomiting, urinary retention, lower limb numbness, motor block, and ecchymosis or hematoma at site of injection will be recorded.
Postoperative Parental satisfaction | 24 hours post-operatively
  Parental satisfaction score will be determined 24 h after the surgery by an anesthetist blinded to the study groups. The child's comfort, activity level and the presence or absence of pain will be used to determine the result as 1 (unsatisfied), 2 (satisfied or good), or 3 (very satisfied or excellent)

REFERENCES:
- [Background] Kendigelen P, Tutuncu AC, Emre S, Altindas F, Kaya G. Pudendal Versus Caudal Block in Children Undergoing Hypospadias Surgery: A Randomized Controlled Trial. Reg Anesth Pain Med. 2016 Sep-Oct;41(5):610-5. doi: 10.1097/AAP.0000000000000447. PMID 27501015
- [Background] Yigit D, Ozen V, Kandirici A, Dokucu AI. Ultrasound-guided dorsal penile nerve block is a safe block in hypospadias surgery: A retrospective clinical study. Medicine (Baltimore). 2022 Jul 1;101(26):e29700. doi: 10.1097/MD.0000000000029700. PMID 35777019